CLINICAL TRIAL: NCT02552667
Title: Efficacy and Safety of HCP1102 Capsule : A Randomized, Double-blind, Active-controlled, Multicenter Phase 3 Clinical Trial
Brief Title: Efficacy and Safety of HCP1102 Capsule
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HM-MOLZ-302
Record Dates: First submitted 2015-09-07; First posted 2015-09-17 (Estimated); Last update posted 2015-09-17 (Estimated); Status verified 2015-09

CONDITIONS: Asthma With Allergic Rhinitis
Keywords: Asthma; Allergic rhinitis
MeSH Terms: conditions — Asthma; Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- HCP1102+HGP0711Placebo (Experimental): HCP1102Placebo+HGP0711Placebo(1week) -> HCP1102+HGP0711Placebo(4weeks) Each 1 capsule, once daily
  Interventions: Drug: HCP1102+HGP0711Placebo
- HCP1102Placebo+HGP0711 (Active Comparator): HCP1102Placebo+HGP0711Placebo(1week) -> HCP1102Placebo+HGP0711(4weeks) Each 1 capsule, once daily
  Interventions: Drug: HCP1102Placebo+HGP0711

INTERVENTIONS:
Drug: HCP1102+HGP0711Placebo — Coadministration of HCP1102 with HGP0711 Placebo for 4-week
  Arms: HCP1102+HGP0711Placebo
Drug: HCP1102Placebo+HGP0711 — Coadministration of HCP1102 Placebo with HGP0711 for 4-week
  Arms: HCP1102Placebo+HGP0711

SUMMARY:
Efficacy and safety of HCP1102 capsule : A randomized, double-blind, active-controlled, multicenter phase 3 clinical trial.

ELIGIBILITY:
Inclusion:

* Age≥15
* Mild or moderate asthma patients with allergic rhinitis
* Patient who meet all criteria of rhinitis
* Patients understood the contents and purpose of this trial and signed informed consent form
* Patients who are capable and willing to write subject diary
* Patients who agree with maintain same environment during clinical trials

Exclusion:

* Nonallergic rhinitis
* Severe asthma
* Other pulmonary disease (pulmonary tuberculosis, COPD) except Asthma
* Medical history of hypertrophic cardiomyopathy, cancer, renal disease, Liver disease, cardiovascular disease, respiratory disease, endocrine disorder, CNS disorder that effect safety
* Medical history of gastrointestinal surgery or gastrointestinal disorders that effect drug absorption
* Alcohol abuse or Drug abuse
* Genetic factor of galactose intolerance or Lapp lactase deficiency or glucose-galactose malabsorption
* pregnant or breast-feeding women or men/women of childbearing age that they don't use contraceptives
* Patient who administered other investigational products within 30 days
* Current smoker Judged to be inappropriate for the study by the investigator after reviewing other reasons

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2014-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change of Mean Daytime Nasal Symptom Score | base line, 3-4week(2weeks)

SECONDARY OUTCOMES:
Change of Mean Daytime Nasal Symptom Score | base line, 1-2week(2weeks), 3-4week(2weeks)
Change of Runny nose (Mean Daytime Nasal Symptom Score) | base line, 1-2week(2weeks), 3-4week(2weeks)
Change of Mean Nighttime Nasal Symptom Score | base line, 1-2week(2weeks), 3-4week(2weeks)
Change of Mean Composite Symptom Score | base line, 1-2week(2weeks), 3-4week(2weeks)
Change of sneezing (Mean Daytime Nasal Symptom Score) | base line, 1-2week(2weeks), 3-4week(2weeks)
Change of pruritus (Mean Daytime Nasal Symptom Score) | base line, 1-2week(2weeks), 3-4week(2weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Choon-Sik Park, M.D., Ph.D., Principal Investigator — Soon Chun Hyang University
Locations (1):
- Soon Chun Hyang University Hospital Bucheon, Bucheon-si, Gyunggi -do, South Korea

REFERENCES:
- [Derived] Kim MK, Lee SY, Park HS, Yoon HJ, Kim SH, Cho YJ, Yoo KH, Lee SK, Kim HK, Park JW, Park HW, Chung JH, Choi BW, Lee BJ, Chang YS, Jo EJ, Lee SY, Cho YS, Jee YK, Lee JM, Jung J, Park CS. A Randomized, Multicenter, Double-blind, Phase III Study to Evaluate the Efficacy on Allergic Rhinitis and Safety of a Combination Therapy of Montelukast and Levocetirizine in Patients With Asthma and Allergic Rhinitis. Clin Ther. 2018 Jul;40(7):1096-1107.e1. doi: 10.1016/j.clinthera.2018.04.021. Epub 2018 Jun 24. PMID 29945738